CLINICAL TRIAL: NCT04152135
Title: Evaluation of Volume Status by Passive Leg Removal Maneuver and Vena Cava Inferior Diameter Measurements Before the Position of Patients in Arthroscopic Shoulder Surgery
Brief Title: Hemodynamic Changes With Passive Leg Raising Maneuver in Patients Undergoing Arthroscopic Shoulder Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, merve namlı emlek, research assistant, Diskapi Teaching and Research Hospital
Other Study IDs: 1
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: passive leg raising maneuver, vena cava inferior diameter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vena cava inferior diameter measurement — Ultrasound equipment with convex probe will be used to measure IVC diameters of the patients in supine position.The IVC sagittal section is described with the probe in the area of subxiphoid. IVC diameters at the junction point of the IVC and right atrium (2cm caudal) are standardized measurement.

SUMMARY:
After intubation of the patients who are undergoing arthroscopic shoulder surgery, plethysmographic waveform will be recorded with blood pressure, heart rate and end-tidal carbon dioxide values and inferior vena cava (IVC) diameter will be measured by ultrasound. New hemodynamic values will be measured after passive leg raising maneuver. Blood pressure, heart rate, end-tidal carbon dioxide values will be re-measured and plethysmographic waveform will be recorded after beach chair position for surgery.

DETAILED DESCRIPTION:
Patients aged between 18-65 years who are undergoing arthroscopic shoulder surgery will be examined. After giving detailed information, voluntary certificate will be taken from patients who accept to participate in the study. Heart rate, oxygen saturation and blood pressure values will be recorded by routine monitoring. After intubation of the patients, plethysmographic waveform will be recorded with blood pressure, heart rate and end-tidal carbon dioxide values and IVC diameter will be measured by ultrasound. New hemodynamic values will be measured after passive leg raising maneuver. Blood pressure, heart rate, end-tidal carbon dioxide values will be re-measured and plethysmographic waveform will be recorded after beach chair position for surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old patients,
* The American Society of Anesthesiologists (ASA) physical status classification score 1-2,
* Patients scheduled for arthroscopic shoulder surgery, intubated, sitting position

Exclusion Criteria:

* Patient refusal,
* Patients with current heart and valve disease,
* Patients with ASA 3-4 status,
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: ASA 1-2 status patients between the ages of 18-65 to be performed arthroscopic shoulder surgery with informed consent
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-29 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
passive leg raising maneuver | 2 minutes
  Head of bed at 0 degrees flat and both legs elevated to 45 degrees
vena cava inferior diameter | 2 minutes
  Ultrasound equipment with convex probe will be used to measure IVC diameters of the patients in supine position.The IVC sagittal section is described with the probe in the area of subxiphoid. IVC diameters at the junction point of the IVC and right atrium (2cm caudal) are standardized measurement.

SECONDARY OUTCOMES:
Blood pressure | 2 minutes
  non-invasive measurement, routine monitoring
Heart rate | 2 minutes
  Routine monitoring
End-tidal CO2 | 2 minutes
  Routine monitoring after intubation
plethysmographic waveform | 2 minutes
  Routine monitoring